CLINICAL TRIAL: NCT05108012
Title: The Safety Evaluation of Ex Vivo Activated Haploidentical Natural Killer Cells (NK) in Recurrent Glioblastoma Multiform Patients (Clinical Trial Phase I)
Brief Title: Nk Cell Therapy for Recurrent Glioblastoma Multiform Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royan Institute (Other Government)
Collaborators: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMB1
Record Dates: First submitted 2020-08-18; First posted 2021-11-04 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-10

CONDITIONS: Glioblastoma Multiform; Recurrent Glioblastoma
Keywords: Natural Killer Cells (NK); Glioblastoma Multiform (GBM)
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: The investigators will enroll 5 patients (3-60 year, both sex, -Lansky performance scale/Karnofsky performance scale: 70-100%) with recurrent Glioblastoma Multiform. A haploidentical donor will enter for each patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Test group (Experimental): The investigators will inject the activated NK cells, 1-3 times with weekly interval into tumor cavity.
  Interventions: Biological: NK cell therapy

INTERVENTIONS:
Biological: NK cell therapy — Activated NK cell injection in tumor cavity of patient with GBM (Glioblastoma Multiform)

SUMMARY:
Glioblastoma multiform is one of the most invasive and deadly cancers that progresses rapidly and leads to death. Surgery with radiotherapy /chemotherapy, as a treatment approach is ineffective in some cases and is associated with relapse and death. Immunotherapy is a special strategy that used as an adjunct therapy in various cancers and among the various methods of immunotherapy; it seems that cell therapy with NK cells is of special importance. A previous study conducted at the Royan Research Institute showed that NK cell proliferation and amplification resulted in the removal of glioblastoma tumor masses in the animal model. The animals had no evidence of tumor recurrence after treatment, and all tumor-related complications resolved after treatment. Therefore, in this study, the investigators intend to evaluate the safety of ex vivo activated cells in 5 patients with glioblastoma multiform whose disease has returned after treatment and who have not had any appropriate treatment.

DETAILED DESCRIPTION:
1- patient selection 2- leukapheresis 3- CD56+ cells isolation 4- NK cells activation 5- assessment of functionality and purity 6- quality control tests 7-NK cell injection in tumor cavity.

ELIGIBILITY:
Age: 3-60 Year -

* Sex: Both
* Lansky performance scale/Karnofsky performance scale: 70-100%
* Life span expectation: >6 months
* Hemoglobin: > 10.0 g/dl
* Platelet count > 100,000/mm³
* Serum total bilirubin < 1.5 times upper limit of normal (ULN)
* ALT and AST < 2.5 times ULN
* Serum creatinine < 1.5 times ULN
* No diagnosis of any other invasive cancer within the past 5 years.
* No concurrent serious medical or psychiatric illness that may interfere with giving informed consent or conducting this study

Exclusion Criteria:

* Patients whose MRI and MRS images is in favor of radio necrosis.
* Due to emergency conditions, the patient cannot tolerate the new treatment
* Lack of a suitable donor or insufficient number of NK cells.
* Development of a new neurological defect after the first injection
* Patient death during surgery
* Closing the reservoir for the next injection (if this problem is resolved, the injections will be done again).

Ages: 3 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Toxicity assay | 4 weeks of last injection
  Toxicity as assessed by NCI CTCAE version 3.0
Adverse Events (AEs) | 1 year
  Defined as the number and severity of adverse events
Safety evaluation | From injection time point up to 48 hours
  Safety evaluated by assessing the medical symptoms measurement: Fever, Hysteria and Convulsion
Safety evaluation | 2 months after injection
  Safety evaluated by assessing the medical symptoms measurement: Meningitis, Neurological disorders
Safety evaluation | From injection time point up to 8 weeks
  Safety evaluated by assessing the medical symptoms measurement: Loss of consciousness
MRI and MRS from the tumor region | 1 months after last dose of NK cell injection up to 1 year each 3 months
  Defined tumoral residua and tumor cell recurrence

SECONDARY OUTCOMES:
Patient survival | After surgery up to an average of 1 year
  Evaluation of patient's life extension followed by NK cell therapy

CONTACTS AND LOCATIONS:
Overall Officials: Niloufar Shayan Asl, MSc, Principal Investigator — Royan Institute for Stem Cell Biology and Technology, ACECR, Tehran, Iran; Monire Mohammad, MSc, Principal Investigator — Royan Institute for Stem Cell Biology and Technology, ACECR, Tehran, Iran; Amirali Hamidieh, MD,PhD, Principal Investigator — Pediatric cell therapy research center, Tehran University of Medical Sciences; Marzieh Ebrahimi, PhD, Study Director — Royan Institute for Stem Cell Biology and Technology, ACECR, Tehran, Iran; Zohreh Habibi, M.D, Study Director — Children's Hospital Medical Center, Tehran University of Medical Science, Tehran, Iran; Abolhossein Shahverdi, PhD, Study Chair — Royan Institute for Reproductive Biomedicine, ACECR, Tehran, Iran
Locations (1):
- Royan institute, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No